CLINICAL TRIAL: NCT00796211
Title: A Single-Center, Randomized, Blinded, Vehicle- Controlled Exploratory Study to Assess the Activity of CRx-197 in Subjects With Plaque Psoriasis
Brief Title: A Single-Center Exploratory Study to Assess the Activity of CRx-197-002 in Plaque Psoriasis
Acronym: 197-002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zalicus (Industry)
Responsible Party: Alka Batycky, Executive Director, Clinical Programs, CombinatoRx
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRx-197-002
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2009-01-15 (Estimated); Status verified 2009-01

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis; CRx-197; nortriptyline; loratadine; CombinatoRx; Dermatology; Erythema; Pruritus
MeSH Terms: conditions — Psoriasis; Erythema; Pruritus | interventions — Nortriptyline; calcipotriene

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): CRx-197 high dose topical cream (0.1% nortriptyline HCl +0.3% loratadine)
  Interventions: Drug: CRx-197
- 2 (Experimental): CRx-197 low dose topical cream (0.1% nortriptyline HCl + 0.1% loratadine)
  Interventions: Drug: CRx-197
- 3 (Active Comparator): 0.1% nortriptyline HCl topical cream
  Interventions: Drug: Nortriptyline
- 4 (Active Comparator): 0.005% calcipotriol topical cream
  Interventions: Drug: Calcipotriol
- 5 (Placebo Comparator): Vehicle of CRx-197 topical cream (placebo)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CRx-197 — CRx-197 high dose topical cream (0.1% nortriptyline HCl +0.3% loratadine)
  Arms: 1
Drug: CRx-197 — CRx-197 low dose topical cream (0.1% nortriptyline HCl + 0.1% loratadine)
  Arms: 2
Drug: Nortriptyline — 0.1% nortriptyline HCl topical cream
  Arms: 3
Drug: Calcipotriol — 0.005% calcipotriol topical cream
  Arms: 4
Other: Placebo — Vehicle of CRx-197 topical cream (placebo)
  Arms: 5

SUMMARY:
This will be a phase 2a single-center, randomized, blinded, vehicle-controlled exploratory study to assess the activity and safety of CRx-197 in subjects with plaque psoriasis. Approximately 20 male or female subjects with chronic plaque type psoriasis, 18 to 70 years of age, will be included in this study.

All subjects with stable psoriatic plaques will receive all of the following treatments each in a separate test field, once each day for four weeks under occlusion:

* CRx-197 high dose topical cream (0.1% nortriptyline HCl +0.3% loratadine)
* CRx-197 low dose topical cream (0.1% nortriptyline HCl + 0.1% loratadine)
* 0.1% nortriptyline HCl topical cream
* 0.005% calcipotriol topical cream
* Vehicle of CRx-197 topical cream (placebo)

ELIGIBILITY:
Inclusion Criteria:

* I01 Subject must voluntarily sign and date the written informed consent prior to any study specific procedures
* I02 Subject must be 18 to 70 years of age
* I03 Subject must have chronic plaque psoriasis and plaque infiltrates of a thickness of a minimum of 150 µm and stable plaques in an area sufficient for up to five test fields and an untreated control field per each plaque
* I04 Subject must be free from a condition/disease that the investigator feels interferes with the interpretation of the study results.
* I05 Females of childbearing potential age should either be surgically sterile (hysterectomy or tubal ligation), or should use a highly effective medically accepted contraceptive regimen.

Exclusion Criteria:

* E01 Erythrodermic, guttate or pustular psoriasis
* E02 Cardiac disease, including recent myocardial infarction, any degree of heart block or other cardiac arrhythmias or valvular heart disease
* E03 Mania or acute delirium or epilepsy
* E04 Narrow angle glaucoma
* E05 Hyperthyroidism by medical history, TSH less than LLN, or a subject receiving thyroid medication
* E06 Diabetes
* E07 Intolerance to lidocaine
* E08 Severe liver disease [ALT laboratory value that exceeds 2.5x ULN]
* E09 Known severe kidney disease, acute urinary retention, prostatic hypertrophy with post void residual urine or laboratory value of creatinine that exceeds 1.5x ULN
* E10 Significant gastrointestinal disease including but not limited to pyloric stenosis or paralytic ileus
* E11 Inflammatory dermatoses except psoriasis; bacterial, viral, or fungal skin infections (at the test plaques); facial rosacea
* E12 Active varicella, tuberculosis, syphilis or post-vaccine reactions
* E13 Autoimmune disease other than plaque psoriasis (e.g., lupus erythematosis)
* E14 Known allergic reactions or hypersensitivity to any of the components of the study treatments
* E15 Allergy to adhesives on the templates used in this study
* E16 UV therapy or significant UV exposure in the four weeks before treatment application
* E17 History of malignancy (except for treated or excised basal cell carcinoma)
* E18 History of drug or alcohol abuse (as defined by the Investigator)
* E19 Symptoms of a clinically significant illness in the four weeks before treatment application that may influence the outcome of the study
* E20 Subject with demonstrated hypercalcemia (calcium greater than ULN) or evidence of Vitamin D toxicity
* E21 Subject with demonstrated hypokalemia (less than LLN)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-11; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by treatment emergent adverse events, physical exams, vital signs, concomitant medications/procedures and subject assessment of pruritus | 6 weeks

SECONDARY OUTCOMES:
Difference in change from baseline in psoriatic infiltrate measured by ultrasound at Days 8, 15, 22, 29 and 43 between CRx-197, nortriptyline, active comparator as well as vehicle of CRx-197 and untreated test field(s) | 6 weeks
Differences in change from baseline in erythema measured by chromametry at Days 8, 15, 22, 29 and 43 between CRx-197, nortriptyline, active comparator, vehicle of CRx-197, untreated test field(s) and normal skin | 6 weeks
Modified PASI at Baseline, and Days 8, 15, 22, 29 and 43 between CRx-197, nortriptyline, active comparator, vehicle of CRx-197, untreated test field(s) | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- ProInnovera, Münster, Germany